CLINICAL TRIAL: NCT01527799
Title: The Physiologic Assessment of Exercise Capacity in Pediatric Sickle Cell Anemia
Brief Title: Exercise Capacity in Pediatric Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert I. Liem, Attending Physician, Hematology, Oncology,Cell Transplantation, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2009-13659; 1K23HL094376 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-07 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell anemia; Exercise testing; Cardiopulmonary disease
MeSH Terms: conditions — Anemia, Sickle Cell; Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma is collected and stored to be analyzed
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with Sickle Cell Anemia: Subjects with Sickle Cell Anemia, 10-21 years of age
- Healthy controls: Healthy controls, 10 to 21 years of age

SUMMARY:
The purpose of this study is to use comprehensive exercise testing to examine causes of exercise limitation in children and young adults with sickle cell anemia.

DETAILED DESCRIPTION:
Although the burden of sickle cell anemia (SCA) on affected individuals is significant, few studies have examined the influence of having SCA on such measures of physical function as exercise capacity. Moreover, the physiologic basis of poor physical functioning in children with SCA is unknown and has not been studied extensively. The purpose of this proposal is to use cardiopulmonary exercise testing (CPET) to gain a comprehensive understanding of exercise capacity, as a measure of physical function, in children and young adults with SCA. The specific aims of this project are to: 1) Measure peak oxygen consumption (VO2), the reference standard for exercise capacity, in children and young adults with SCA classified by primary pathophysiologic contributor to their decreased exercise capacity, and 2) Examine the acute inflammatory response, measured by an increase in soluble vascular cell adhesion molecule (sVCAM) activity, in subjects undergoing CPET. These aims will be performed in 60 subjects with SCA and 30 matched controls without SCA. In a secondary analysis, we will also study the impact of baseline exercise capacity and the inflammatory response to exercise on short and long-term disease related morbidity. This study is essential because it will address several areas of exercise capacity, including the physiologic contributors to exercise limitation that remain fundamental knowledge gaps in SCA.

ELIGIBILITY:
Inclusion Criteria:

1. age 10 to 21 years old; AND
2. Hb SS or S-β0 thalassemia disease, confirmed by hemoglobin analysis

Exclusion Criteria:

1. inability to perform maximal testing due to physical limitation (e.g. stroke or avascular necrosis); OR
2. history of exercise-induced syncope or arrhythmias. Subjects will wait at least 2 weeks following any vaso-occlusive pain episode and 12 weeks following any disease-related complication requiring transfusion support. Individuals on hydroxyurea will be eligible. A total of 30 controls without SCA or sickle cell trait will be matched for age, sex and race and recruited from the siblings, friends or relatives of subjects enrolled on this study

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sickle cell anemia patients followed at Children's Memorial Hospital. Healthy controls without sickle cell anemia are recruited through flyers posted in Children's Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
VO2 max on cardiopulmonary exercise test | Baseline

SECONDARY OUTCOMES:
Skin fold measurements to detemine percent body fat | Baseline
All patient reported pain episodes | Every 2 months up to 2 years after baseline
Change in secondary biomarkers in response to exercise test | Baseline (Pre-exercise) and Post-exercise
Change in VCAM level in response to exercise testing | Baseline (pre-exercise) and Post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Liem, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States